CLINICAL TRIAL: NCT05818735
Title: Efficacy and Safety of Electroacupuncture on Treating the First Episode of Mild to Moderate Depression
Brief Title: Effect of Electroacupuncture on Treating the First-episode Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Municipal Hospital of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Mental Health Center (Other); Xuhui Central Hospital, Shanghai (Other); Shanghai Huangpu District Mental Health Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shifen Xu
Record Dates: First submitted 2023-03-15; First posted 2023-04-19 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Depression
Keywords: first-episode depression; electroacupuncture; anti-depressants; sham acupuncture; placebo drugs; randomized controlled trial
MeSH Terms: conditions — Depression | interventions — Electroacupuncture; Therapeutics; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the electroacupuncture group (Experimental): the electroacupuncture and the placebo drug
  Interventions: Other: electroacupuncture (EA) treatment; Drug: Placebo
- the drug group (Placebo Comparator): the sham acupuncture and the drug Escitalopram
  Interventions: Other: sham acupuncture (SA) treatment; Drug: Escitalopram 10mg

INTERVENTIONS:
Other: electroacupuncture (EA) treatment — The regular acupuncture treatment will be applied at the acupoints including Baihui (GV20), Yintang (GV29), Guanyuan (RN4), Qihai (RN6), bilateral ZuSanli (ST36) and bilateral SanYinjiao (SP6). After needle insertion, rotating or lifting-thrusting manipulation will be applied for 'De qi' sensation. Three pairs of electrodes of the electroacupuncture apparatus will be connected to the needles of GV20 and GV29, and bilateral ST36 and SP6 for 25 minutes, delivering a continuous wave with a frequency of 2-8Hz which is based on the tolerance of each patient. The selection of matching acupuncture points will be determined by the acupuncturist according to the patients' different syndrome patterns.
  Arms: the electroacupuncture group
Other: sham acupuncture (SA) treatment — The sham acpunture treatment will be applied at the same acupoints as the EA treatment with the Streitberger placebo needles. When the blunt needle tip of the placebo needles touches the skin, the patient will get a pricking sensation, but there is no real needle inserted into the skin. The electroacupuncture apparatus will be set on the table beside the patients and two pairs of electrodes will be connected to the needles at bilateral ST36 and SP6. Acupuncturists will turn on the apparatus but all indicators will be set to '0'. Participants will be informed when needles are removed after 25 minutes. Acupuncturists will use dry cotton balls to press the skin around the acupoints when withdrawing the needles so that patients can feel the withdrawal of the 'needles'.
  Arms: the drug group
Drug: Escitalopram 10mg — Escitalopram will be used as the antidepressants for relieving patients' depressive mood. The dose of the drug will be the minimum clinical starting dose of 10 mg once daily, taken orally in the morning, for a period of 3 months. During the intervention period, patients will be allowed to increase the drug dose (up to 20 mg) according to their mental status. Patients will record the details of the drug dose, duration of dosing,responses and possible side effects on a drug dairy. Pateints will receive 7 tablets of escitalopram from an independent dispencer at a set time each week. They may receive additional dose of escitalopram once again during the week if necessary and it will be recorded by the dispenser.
  Other Names: real drug application
  Arms: the drug group
Drug: Placebo — Placebo drugs are tablets of the same color and size as escitalopram tablets, consisting mainly of starch, and will be tested for safety before being used in the trial. The way the medication is dispensed, the details of how the medication is administered, the dosage, and the record of the drug diary are consistent with the application of the real drugs.
  Other Names: placebo drug application
  Arms: the electroacupuncture group

SUMMARY:
Depression is a disease that endangers the physical and mental health of all human beings. Only 30-40% of patients with initial episode depression are cured after treatment with antidepressants. Acupuncture is a widely recognized therapy to treat depression in clinical practice, and it can effectively relieve the depressive mood and improve related physical symtoms in patients with mild to moderate depression. This randomised controlled trial (RCT) is aimed to investigate the efficacy and safety of electroacupuncture (EA) in the treatment for patients with the first-episode of mild to moderate depression.

DETAILED DESCRIPTION:
Patients will be recruited from the outpatient clinics in Shanghai Municipal Hospital and Shanghai Mental Health Center by Wechat and posters. A total of 204 eligible patients will be randomly allocated to two groups by a randomized block design: the electroacupuncture (EA) group (receiving EA treatment and taking the placebo drugs), and the antidepressants group (receiving sham acupuncture and taking the escitalopram ). After a one-week baseline evalauation, participants will enter a 9-month observation period in this trial, with a 3-month intervention period and a 6-month follow-up period. The interventiuon period will last for 12 weeks, with 3 sessions of real or sham acupuncture treatment per week for the first 8 weeks, and 2 sessions per week for the remaining 4 weeks. The escitalopram or the placebo will be given to the patients at a set time once a week during the 12-week intervention period, with daily oral dose of 10mg or up to 20mg as the maximum dose. Excperts in the Shanghai Mental Health Center will help the participants to adjust the drug dosage during the intervention period. The primary outcome is the 17-item Hamilton Rating Depression Sclae (HRDS-17) at week 12. The secondary outcomes include the recovery rate and the remission rate of depression, the Patient Health Questionnaire(PHQ-9) and the Medical Outcomes Study 36-Item Short Form (SF-36). Adverse effects will be assessed by the Treatment Emergent Symptom Scale through the trial. The software SPSS Version 24.0 for Windows will be used to do the data analysis. All statistical analyses will be based on the intention-to-treat (ITT) population of all randomly assigned patients, with a 2-sided significance level of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who meet the diagnostic criteria of depression according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition.
2. Participants whose HDRS-17 score is 17-25 (mild-to-moderate depression).
3. Participants who suffer from depression for the first time.
4. Patients who have not taken any previous antidepressants.
5. Patients who are assessed as low risk for suicide.
6. Participants who have not received acupuncture treatment for at least 1 year.
7. Participants who voluntarily agree with the investigation and sign a written informed consent form.

Exclusion Criteria:

1. Participants with secondary depressive disorders caused by organic diseases, medicine or psychotic disorders.
2. Participants who are in the depressive episode of bipolar disorder, or suffering from dysthymia, reactive depression and depressive syndrome caused by other diseases.
3. Participants who had severe organic brain diseases and other serious physical diseases.
4. Participants with a history of alcohol abuse or drug dependence.
5. Participants who have enrolled in other clinical trial within 1 months.
6. Pregnant or lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
17-item Hamilton Depression Rating Scale (HDRS-17) | Week 12
  The HDRS-17 is an observer-rating questionnaire with 17 items used to assess the symptoms of patients diagnosed as suffering from depressive states. Each item is rated in 3-point or 5-point scales. A higher total score indicates a higher depression level.

SECONDARY OUTCOMES:
Recovery rate of depression | Week 12
  the percentage of patients with an HDRS-17 score ≤8
Remission rate of depression | Week 12
  the percentage of patients' HDRS-17 score between 8 and 12
HDRS-17 | Week 4, week 8, week 16, week 24 and week 36
  The HDRS-17 is an observer-rating questionnaire with 17 items used to assess the symptoms of patients diagnosed as suffering from depressive states. Each item is rated in 3-point or 5-point scales. A higher total score indicates a higher depression level.
Patient Health Questionnaire(PHQ-9) | Week 4, week 8, week 16, week 24 and week 36
  The PHQ-9 is developed according to the American Diagnostic Criteria for Major Depressive Disorder and is recommended by the WHO as an important tool for screening and assessing the depressive status of patients. It consists of 9 items that are easily and effectively used to understand a subject's depression. The higher the total score indicates the more severe depression.
The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) | Week 4, week 8 and week 12
  It is one of the most widely used quality-of-life assessment scales with good reliability and validity. It provides a comprehensive overview of the participants' level of quality of life in eight dimensions: physiological functioning, physical functioning, somatic pain, general health status, energy, social functioning, emotional functioning, and mental health. A combination of item response(s) is then aggregated to calculate a score for each of the eight dimensions. The scores for each dimension range from 0 to 100, with higher scores indicating better health status.
Drug dairy | Up to 12 weeks
  A drug record booklet will be issued by the study staff to each patients, and the participants will be asked to record the actual dose, frequency, time of taking drug or side effects everyday.
Adverse events（AEs） | Up to 12 weeks
  Adverse events (AEs) in the trial includes any abnormal events and all types of medical events that were clearly or suspected to be related to the real and sham acupuncture treatment or the drug. Patients may occur focal skin infections, subcutaneous hematomas, and dizziness during the acupuncture treatment, or exacerbation of the condition due to excessive treatment stimulation. AEs including sedation, dizziness, sleep disorders, or constipation due to the drug will be recorded as well. Cold, trauma, or other medical events that resulted in hospitalization during the trial will be also included as AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Shifen Xu, Doctor, Principal Investigator — Shanghai Municipal Hospital of Traditioal Chinese Medicine
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Results will be published by the investigators in academic journals. Data obtained through this study will be provided to qualified researchers with academic interest in acupucnture treatment for depression. Data or samples shared will be coded. The IPD can be shared by sending email to the PI Shifen Xu (xu_teacher2006@126.com) .
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and SAP and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact Shifen Xu.